CLINICAL TRIAL: NCT00442442
Title: Clinical Evaluation of Mosquito Coils to Control Malaria in China
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Yunnan Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IDCVNHIL01; LSHTM ITDCVP89
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Malaria
Keywords: Malaria; mosquito control; mosquito coils; LLIN
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): No treatment control
- 2 (Active Comparator): LLIN Nets
  Interventions: Device: LLIN
- 3 (Experimental): Mosquito Coils
  Interventions: Device: mosquito coils
- 4 (Experimental): Mosquito coils & LLIN
  Interventions: Device: mosquito coils

INTERVENTIONS:
Device: mosquito coils — mosquito coil / night mosquito coil & LLIN / night
  Arms: 3; 4
Device: LLIN — Sleep under LLIN every night
  Arms: 2

SUMMARY:
Although mosquito coils are widely used, there is no robust evidence that their use can provide clinical reduction in malaria. This study will randomise 4 groups of 400 houses, each with 5 people, in rural China and monitor cases of malaria in each group each month for 6 months. The treatment groups will include Coils, Treated bed nets, Coils plus treated bed nets, or no treatment (control). All cases detected will be given prompt appropriate treatment.

DETAILED DESCRIPTION:
Mosquito coils are extremely widely used by households across the world and reportedly make up the largest single family expenditure on any health-related items in many developing Countries. Despite their widespread use there has been no robust clinical evaluation to determine whether they can provide protection from malaria. This study is designed to determine if using coils (and / or LLIN) each evening can reduce malaria at the household level.

The study will be a single-blind, randomised clinical evaluation clustered at the household level. There will be 4 treatment arms, Coils / Insecticide treated nets / Coils + ITN / No treatment. Each arm will include 400 households each with 5 people / household (total of 8000 people). A maximum of 20% of houses in any village will be enrolled to reduce any effects of diversion of mosquitoes by any treatment. Epidemiological factors and baseline malaria prevalence will be recorded during a pre-intervention baseline month by questionnaire and rapid diagnostic test (RDT) using species-specific dip sticks for malaria. Post intervention will be 5 further monthly visits during the malaria season to detect new cases by RDT, reported fevers and operational data (compliance, adverse effects etc). Primary outcome clinical measures will be incidence of malaria (P. falciparum / P. vivax) comparing new cases in each of the 3 treatment & non-treatment groups. All cases will be treated promptly according to local policy. At the end of the study, all households which did not have a treated bed net will be provided with one.

Secondary non-clinical outcome measures will include entomological data collected in houses using / non using coils in sentinel villages at baseline & during the study. CDC mosquito light traps will be used to record number / species / feeding status / parity (age) / sporozoite infection rates of mosquitoes in houses using / not-using coils following a randomised latin square design. Such entomological data can be used to determine reduction in vector species mosquitoes entering houses using coils and / or ITN.

Ethical approval for the study has been granted by the LSHTM University of London Ethics Committee and the Yunnan Bureau of Health, P.R.China.

ELIGIBILITY:
Inclusion Criteria:

* 6 years plus,
* No allergy to products in use,
* Not pregnant / breast feeding

Exclusion Criteria:

* Not sleeping at home each night

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2007-04; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Malaria cases | 6 months

SECONDARY OUTCOMES:
Fever reports | 6 months
User acceptance | 6 months
entomological data | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hill, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Hong Ning Zhou, MSc, Principal Investigator — Yunnan Institute of Parasitic Diseases
Locations (1):
- Yunnan Institute of Parasitic Diseases, Pu'er, Yunnan, China

REFERENCES:
- [Derived] Hill N, Zhou HN, Wang P, Guo X, Carneiro I, Moore SJ. A household randomized, controlled trial of the efficacy of 0.03% transfluthrin coils alone and in combination with long-lasting insecticidal nets on the incidence of Plasmodium falciparum and Plasmodium vivax malaria in Western Yunnan Province, China. Malar J. 2014 May 31;13:208. doi: 10.1186/1475-2875-13-208. PMID 24885993